CLINICAL TRIAL: NCT02009384
Title: A Phase II Open-Label Study of Ipilimumab Administered to Stage IIIC and Stage IV Melanoma Patients After Regulatory T Cell Depletion With Denileukin Diftitox
Brief Title: Ipilimumab Administered to Stage IIIC Stage IV Melanoma After Reg. T Cell Depletion With Denileukin Diftitox
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment r/t requirement of prior treatment with denileukin diftitox
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Jason Chesney, Director, James Graham Brown Cancer Center, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-MEL-11-01
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab (Experimental): IV ipilimumab
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — administration of IV ipilimumab for up to 4 cycles

SUMMARY:
This is an open-label, clinical efficacy study of Ipilimumab in patients with Stage IIIC and Stage IV melanoma who have recently been treated with Denileukin Diftitox. Approximately 42 patients with radiographically measurable melanoma who have received at least one cycle of Denileukin Diftitox will be enrolled and treated in the study.

DETAILED DESCRIPTION:
This is an open-label, clinical efficacy study of Ipilimumab in patients with Stage IIIC and Stage IV melanoma who have recently been treated with Denileukin Diftitox. Approximately 42 patients with radiographically measurable melanoma who have received at least one cycle of Denileukin Diftitox will be enrolled and treated in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age;
2. Patients with histological confirmed melanoma (Stage IIIC or Stage IV, American Joint Commission on Cancer);
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2;
4. Life expectancy ≥3 months;
5. Treatment with Denileukin Diftitox within 42 days prior to first dose of Ipilimumab;
6. At least 1 site of radiographically measurable disease by immune-related response criteria (irRC);
7. Adequate hematologic, renal, and liver function as defined by laboratory values performed within 42 days prior to initiation of dosing:

   * Absolute neutrophil count (ANC) ≥1.0 x 109/L;
   * Platelet count ≥100 x 109/L;
   * Hemoglobin ≥8 g/dL;
   * Serum creatinine ≤3 x upper limit of normal (ULN)
   * Total serum bilirubin ≤2 x ULN;
   * Serum aspartate transaminase (AST/SGOT) or serum alanine transaminase (ALT/SGPT) ≤2x ULN, and ≤3 x ULN if liver metastases are present.
8. Fertile males should use an effective method of contraception during treatment and for at least 3 months after completion of treatment, as directed by their physician;
9. Pre-menopausal females and females <2 years after the onset of menopause should have a negative pregnancy test at Screening. Pre-menopausal females must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 90 days after the last dose of study drug. Females of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year;
10. Before study entry, written informed consent must be obtained from the patient prior to performing any study-related procedures.

Exclusion Criteria:

1. Prior treatment with Ipilimumab;
2. Known hypersensitivity to Ipilimumab or any of its components;
3. Steroids within one week prior to initiation of Ipilimumab.
4. Pre-existing autoimmune colitis.
5. Patients with an allograft requiring immunosuppression;
6. Known positive human immunodeficiency virus (HIV)
7. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives, or avoidance of pregnancy measures;
8. Have any other uncontrolled infection or medical condition that could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chesney, MD, Principal Investigator — Brown Cancer Center, University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was Terminated due to low subject enrollment [r/t requirement of prior treatment with denileukin diftitox] Data was not analyzed
Pre-assignment Details: Study was Terminated
Groups:
- Ipilimumab: IV ipilimumab
  Ipilimumab: administration of IV ipilimumab for up to 4 cycles
  Study was Terminated due to low subject enrollment [r/t requirement of prior treatment with denileukin diftitox] Data was not analyzed
Period: Overall Study
Arm/Group | Ipilimumab
Started | 2 (Study was Terminated due to low subject enrollment Data was not analyzed)
Completed | 0 (Study was Terminated due to low subject enrollment Data was not analyzed)
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants] — Age at Baseline
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] — Age collected by medical record
  years | 67 [65 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — collected by medical record
  Participants
    Female | 0
    Male | 2
Region of Enrollment [Number; unit: participants] — based on subject address
  participants
    United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Using Immune-related Response Criteria (irRC)
Description: no outcomes available, Study was Terminated due to low subject enrollment [r/t requirement of prior treatment with denileukin diftitox] Data was not analyzed
Time Frame: baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Population: no outcomes available, Study was Terminated due to low subject enrollment [r/t requirement of prior treatment with denileukin diftitox] Data was not analyzed
Arm/Group | Ipilimumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All AEs During study treatment and 21 days following end of treatment will be documented and reported if applicable. Adverse events occurring between the time of signing informed consent to the date of the first dose will NOT be captured as AEs unless the AE is a direct result of a study-specific procedure or results in death from an event other than PD
Groups:
- Ipilimumab: dosage:3 mg/kg of subject weight dosage form: Intravenous administration on Ipilimumab frequency of administration: Ipilimumab: administration of IV ipilimumab every three weeks for up to 4 cycles
Arm/Group | Ipilimumab
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab (N=2)
Grade: 3 Encephalopathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes